CLINICAL TRIAL: NCT04344496
Title: The Cancer Genome Atlas and Recurrence Risk Prediction of East Asian Breast Cancer: a Multicenter Collaborative Study
Brief Title: East Asian Breast Cancer Genome Atlas and Recurrence Risk Prediction
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805027RSA
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PAM50 — PAM50 results is as one of the references for the physicians and the participants to choose adjuvant treatments.

SUMMARY:
This project aims to establish the cancer genome atlas and the platform of recurrence risk prediction specific for East Asian breast cancer patients. The study was planned to collect blood sample, fresh tumor tissue, and paraffin embedded tumor tissue from 2000 patients. Aims to identify unique genetic alterations in Asian tumors, to identify the susceptible genes for breast carcinogenesis in East Asia, and to establish the new platform for accurate prediction of recurrence. The investigator will explore the association of patient outcomes with the genetic alterations from the cancer atlas of East Asian breast tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged more than 20-year-old at the time of informed consent.
* 2. An unconfirmed breast tumor, or have histologically confirmed invasive breast cancer.
* 3. Have radiological or objective evidence of breast tumor size ≥1 cm.
* 4. Be able to comply with study procedures to collect the clinical medical information, blood sample, fresh tumor tissue, and 12 sections of paraffin embedded tumor tissue.
* 5. Be able to sign an informed consent.

Exclusion Criteria:

* 1. Have histologically confirmed ductal carcinoma in situ (DCIS).
* 2. Stage I, II or III breast cancer patients who have received neoadjuvant treatments, including chemotherapy, hormonal therapy, or targeted therapy.
* 3. Stage IV or metastatic breast cancer patients who have received chemotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I, II, III or IV Breast Cancer
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of unique genetic alterations | 3 years
  To establish the cancer genome atlas and identify the susceptible genes for breast carcinogenesis in East Asia

SECONDARY OUTCOMES:
Recurrence rate | 10 years
  To establish the new platform for accurate prediction of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan